CLINICAL TRIAL: NCT03902314
Title: Lidocaine Infusions for Children Undergoing Combined Tonsillectomy and Adenoidectomy: A Double-Blinded, Randomized, Placebo-Controlled Trial
Brief Title: Lidocaine Infusion for Pain Relief in Children Scheduled for Tonsillectomy and Adenoidectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Edward Suh MD, Principal Investigator; Clinical Instructor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 014118
Record Dates: First submitted 2019-03-27; First posted 2019-04-04 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Children, Only; Tonsillar Hypertrophy; Adenoid Hypertrophy
Keywords: Lidocaine; Tonsillectomy and Adenoidectomy; Pain
MeSH Terms: conditions — Pain | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomly assigned into one of two intervention groups:
  Group 1: systemic lidocaine infusion Group 2: normal saline infusion
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Anesthesia care providers will be acquiring the study solution from the institution's pharmacy (lidocaine or saline) to administer perioperatively. The pharmacy will prepare the study solutions per randomization and label the solution as the study solution without reference to lidocaine or saline. Per protocol, the care providers will then administer the study solution as a weight based infusion.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Active Comparator): Lidocaine infusion at 2 mg/kg/hr will be started in the operating room and continue in the recovery period for 60 minutes.
  Interventions: Drug: Lidocaine Iv
- Saline (Placebo Comparator): Saline infusion at 2 mg/kg/hr will be started in the operating room and continue in the recovery period for 60 minutes.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Lidocaine Iv — Intravenous infusion
  Arms: Lidocaine
Drug: Saline Solution — Intravenous infusion
  Arms: Saline

SUMMARY:
Lidocaine is widely available and is a very commonly used local anesthetic. When administered intravenously, lidocaine infusions have anti-inflammatory effects and have significantly decreased the reliance on opioid use for adequate pain management in adult abdominal and spine surgeries. A major advantage of lidocaine infusion is that it is not associated with a significant side effect profile.The role of lidocaine in pediatric acute perioperative pain remains limited.

DETAILED DESCRIPTION:
The aim of the study is to determine if using lidocaine continuously during anesthesia care will decrease post-operative pain for children having their tonsils and adenoids removed.

ELIGIBILITY:
Inclusion Criteria:

- scheduled tonsillectomy and adenoidectomy with or without myringotomy/PE tubes at Hasbro Children's Hospital

Exclusion Criteria:

* history of allergies to local anesthetics
* physical or developmental delays
* psychiatric illness
* current use of sedative or anticonvulsive medications
* use of premedication (oral/nasal)
* pre-existing cardiovascular, renal, or hepatic disease
* pre-existing cerebral or neuromuscular disease
* patient with personal or family history of malignant hyperthermia
* recent history of upper respiratory infection within last 7 days
* regular use of analgesic medications

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Change in Pain Scores | 15 minute intervals in postanesthesia care unit; up to 120 minutes following surgery.
  FLACC scale includes 5 categories (Face, Legs, Activity, Cry, Consolability) of pain behaviors scored from 0-2 to provide a total pain score ranging from 0 to 10 with higher numbers indicating greater or worse pain.

SECONDARY OUTCOMES:
Opioid consumption | Total perioperative period: time in the operating room until time of discharge to home from the postoperative anesthesia care unit (PACU)
  Morphine equivalents
Emergence delirium scores | 5 minute intervals for the first 30 minutes in postanesthesia care unit, then every 15 minutes for an additional 90 minutes after surgery
  Pediatric Anesthesia Emergence Delirium (PAED) scale to differentiate emergence delirium from postoperative pain. The scale includes 5 categories (eye contact, purposefulness of actions, awareness of surroundings, restlessness, inconsolable) each scored from 0 to 4 to provide a total score ranging from 0 to 20 with higher numbers being worse indicating that the emergence behaviors correlate better with emergence delirium.
Parental satisfaction with the anesthetic | Evaluated once on postoperative day 1 (or 24 hours after surgery)
  Measured on a scale from 0 to 10, where 0 means very unsatisfied and 10 means very satisfied; higher numbers are better

CONTACTS AND LOCATIONS:
Overall Officials: Edward Suh, MD, Principal Investigator — Lifespan
Locations (1):
- Hasbro Children's Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guntinas-Lichius O, Volk GF, Geissler K, Komann M, Meissner W. Pain after pediatric otorhinolaryngologic surgery: a prospective multi-center trial. Eur Arch Otorhinolaryngol. 2014 Jul;271(7):2049-60. doi: 10.1007/s00405-014-2914-9. Epub 2014 Feb 9. PMID 24510234
- [Background] Howard D, Davis KF, Phillips E, Ryan E, Scalford D, Flynn-Roth R, Ely E. Pain management for pediatric tonsillectomy: an integrative review through the perioperative and home experience. J Spec Pediatr Nurs. 2014 Jan;19(1):5-16. doi: 10.1111/jspn.12048. Epub 2013 Aug 21. PMID 24393224
- [Background] Koppert W, Ostermeier N, Sittl R, Weidner C, Schmelz M. Low-dose lidocaine reduces secondary hyperalgesia by a central mode of action. Pain. 2000 Mar;85(1-2):217-24. doi: 10.1016/s0304-3959(99)00268-7. PMID 10692621
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107